CLINICAL TRIAL: NCT03924102
Title: Cardiac Perfusion and Metabolism With [11C] Acetate PET/CT is Associated With Hematopoietic System Activation in Acute Decompensated Heart Failure: An Imaging Sub-study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was not able to enroll any eligible subjects.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pradeep Bhambhvani, MD, Professor, Division of Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R19-056
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Metabolism

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- patients with acute decompensated systolic and diastolic heart (Experimental)
  Interventions: Drug: Cardiac Perfusion and Metabolism with [11C] Acetate PET/CT

INTERVENTIONS:
Drug: Cardiac Perfusion and Metabolism with [11C] Acetate PET/CT — A rest and stress imaging study will be conducted on the PET/CT scanner with [11C] Acetate.

SUMMARY:
The purpose of this sub-study is to use positron emission tomography and computed tomography imaging (PET/CT) with an investigational drug called [11C] acetate to see if inflammation in patients with acute decompensated heart failure (ADHF) can cause changes in blood flow and oxygen use in the heart. This study may help physicians better understand how to treat patients diagnosed with ADHF in the future.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Enrollment in the UAB CMC-ADHF study under the separate UAB approved research protocol (IRB-300000114, PI Rajapreyar)
* Negative urine or serum β-hCG test within 48 hours of [11C] acetate administration in women of child bearing potential. Women who are post-menopausal with at least 1 year since last menses or documented surgical sterilization will not require pregnancy testing.

Exclusion Criteria:

* Inability to provide informed consent
* Pregnancy
* Inability to lie still for the imaging study
* Weight exceeding the weight limit of the PET imaging table (500 pounds).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Inflammation in patients with acute decompensated heart failure (ADHF) will be measured with rest-stress [11C] acetate PET/CT to see if the inflammation can cause changes in the blood flow and oxygen use in the heart. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States